CLINICAL TRIAL: NCT06208748
Title: A Phase II Trial of Bezuclastinib in Combination With Sunitinib in Patients With GIST Who Progressed on Sunitinib Monotherapy
Brief Title: SARC044: A Phase II Trial of Bezuclastinib in Combination With Sunitinib in Patients With GIST
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Cogent Biosciences, Inc. (Industry); Dana-Farber Cancer Institute (Other); The Life Raft Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC044
Record Dates: First submitted 2023-12-20; First posted 2024-01-17 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Gastrointestinal Stromal Tumors; GIST
Keywords: GIST; Gastrointestinal Stromal Tumors; Sarcoma; Sunitinib; Bezuclastinib; exon 11 or exon 9 primary KIT mutation
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma | interventions — Sunitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- bezuclastinib in combination with sunitinib (Experimental): Bezuclastinib 600 mg (tablet) administered orally daily Sunitinib 37.5 mg administered orally daily
  Patients will begin bezuclastinib and add sunitinib 2 weeks later. Each cycle is 28 days.
  Interventions: Drug: Bezuclastinib in combination with sunitinib

INTERVENTIONS:
Drug: Bezuclastinib in combination with sunitinib — Bezuclastinib in combination with sunitinib (sutent)

SUMMARY:
This is an open label, single arm, phase 2 trial investigating bezuclastinib plus sunitinib in patients with GIST who have previously progressed on sunitinib.

DETAILED DESCRIPTION:
This is an open label, single arm, phase 2 trial investigating bezuclastinib plus sunitinib in patients with GIST who have previously progressed on sunitinib. After washout, patients will begin bezuclastinib and add sunitinib 2 weeks later. Patients will continue on treatment until progression, unacceptable toxicity, or withdrawal of consent. Patients may stay on treatment beyond progression if there is clinical benefit in the opinion of the investigator. Imaging response assessments will be performed every 8 weeks until the participant reaches 15 months on study. After 15 months, response assessments may be performed every 3 months. Circulating tumor DNA (ctDNA) will be collected at baseline, with sequential initiation of bezuclastinib and sunitinib, at the first response assessment, and at the time of progression. In a subset of 20 patients, PET/CT will be performed at baseline and with sequential initiation of bezuclastinib and sunitinib, and tumor biopsies will be performed on cycle 2 day 1 for correlative studies. EORTC QLQ-C30 will be administered during the study to assess patient-reported quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age minimum of 18 years
* Histologically confirmed, inoperable or metastatic GIST with an exon 11 or exon 9 primary KIT mutation. Other primary KIT mutations (e.g., exon 13, exon 17) will be considered on a case-by-case basis after discussion with the Principal Investigator. Pathology reports including mutational analysis should be available for review by the Sponsor.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2 (See Appendix A).
* Prior progression on or intolerance to imatinib. Imatinib intolerance is defined as discontinuation of imatinib due to an adverse event(s) related to treatment with imatinib that was not manageable with dose modifications.
* Documented disease progression on sunitinib of at least 25 mg daily as continuous treatment, or 37.5 mg daily with the 4 weeks on/2 weeks of schedule.
* At least one site of measurable disease on CT/MRI scan as defined by modified RECIST version 1.1 (mRECIST v1.1) criteria.
* Resolution of toxicities from prior therapy to ≤Grade 1 (or baseline), including clinically significant laboratory abnormalities, prior to the first dose of the study drug.
* Adequate organ function:
* Absolute Neutrophil Count (ANC) ≥ 1 x 109/L (unsupported for 7 days, or 14 days if pegfilgrastim was administered)
* Platelets ≥ 100 x 109/L (unsupported for 14 days)
* Hemoglobin ≥8 g/dL (unsupported for 14 days)
* ALT and AST ≤ 2.5 x institutional upper limit of normal (ULN) or ≤ 5.0 x institutional ULN in the presence of hepatic metastases.
* Serum bilirubin ≤ 1.5 x institutional ULN. NOTE: Patients with elevated bilirubin secondary to Gilbert's disease are eligible to participate in the study provided that direct bilirubin ≤1.5 x institutional ULN and indirect bilirubin ≤3 x institutional ULN
* Estimated glomerular filtration rate ≥45 mL/min/1.73 m2
* Ability and willingness to provide written, voluntary informed consent
* Ability to swallow pills
* For male subjects, unless having undergone permanent sterilization (includes bilateral orchidectomy), agreement to use effective barrier contraception (i.e., condoms) during the study treatment period and for 6 weeks after the last dose of study drug.
* For women of childbearing potential (WOCBP), confirmation of negative serum or urine pregnancy test prior to dosing with the study drug and agreement to the use of highly effective method of contraception with or without a barrier contraception method during the study treatment period and for 6 weeks after the last dose of the study drug. Female subjects who are using hormonal contraception must agree to remain on a stable regimen throughout the study unless a change is deemed medically necessary by the Investigator.

WOCBP are defined as defined as physiologically and anatomically capable of becoming pregnant, unless they meet one of the following conditions:

* Postmenopausal: 12 months of natural (spontaneous) amenorrhea without an alternative medical cause
* Prior hysterectomy
* Prior bilateral oophorectomy
* Prior bilateral salpingectomy

Highly effective methods of birth control includes:

* Combined (estrogen- and progesterone-containing) hormonal contraception associated with inhibition of ovulation, delivered orally, intravaginally, or transdermally
* Progestogen-only hormonal contraception associated with inhibition of ovulation, delivered orally, via injection, or implanted
* An intrauterine device (IUD)
* An intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized partner - provided the partner is the sole sexual partner of the WOCBP study participant and that the vasectomized partner has received medical assessment of the surgical success
* Sexual abstinence, when consistent with the preferred and usual lifestyle of the subject, can be considered acceptable based on the evaluation of the Investigator, who should take into consideration the duration of the clinical study. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation) and withdrawal are not considered acceptable methods of contraception.

  * Life expectancy of > 12 weeks
  * For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. For participants with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
  * Patients with central nervous system disease are eligible for enrollment if they have received prior radiotherapy or surgery to sites of CNS metastatic disease and are without evidence of clinical or radiographic progression at the time of enrollment.

Exclusion Criteria:

* Prior exposure to bezuclastinib.
* Prior anticancer drug less than 5 half-lives of the parent drug and/or its active metabolite(s) or 14 days (whichever is shorter) prior to the first dose of the study drug.
* Received strong CYP3A4 inhibitor(s) or inducer(s) within 14 days or 5 drug half-lives before the first dose of the study drug, whichever is longer, or the need to continue treatment with strong CYP3A4 inhibitor(s) or inducer(s) during the study.
* GIST without primary activating mutations in KIT exons 11 or 9. Other primary KIT activating mutations will be considered on a case-by-case basis. Patients with GIST with other mutations (e.g., PDGFRA, SDHx, BRAF, or NF1) or unknown genotype are excluded.
* Known or suspected hypersensitivity to bezuclastinib or sunitinib and their components.
* Unacceptable toxicity with prior sunitinib at 25 mg daily.
* Clinically significant cardiac disease, defined by any of the following:
* Clinically significant cardiac arrhythmias and/or the need for antiarrhythmic therapy (excluding beta blockers or digoxin). Subjects with controlled atrial fibrillation are not excluded.
* Congenital long QT syndrome or use of concomitant medications known to prolong the QT interval as defined in Appendix D.
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >470 milliseconds [ms] using Fridericia's QT correction formula).
* Clinically significant history of cardiac disease or congestive heart failure >New York Heart Association Class II. Subjects must not have unstable angina (anginal symptoms at rest) or new-onset angina within 3 months or myocardial infarction within 6 months prior to enrollment.
* Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis, or pulmonary embolism within the 6 months before study drug initiation (except for adequately treated catheter-related venous thrombosis occurring more than 1 month before the first dose of study drug).
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen may be included after discussion with the Principal Investigator.
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol.
* Patients known to be seropositive for human immunodeficiency virus (HIV) 1 or 2. HIV testing is not required as part of screening.
* Major surgery (including abdominal laparotomy) within 4 weeks prior to the first dose of study drug, or subjects who have not recovered adequately from prior surgery.
* Gastrointestinal abnormalities including, but not limited to, significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption
* Any active bleeding, excluding hemorrhoidal or gum bleeding
* Women who are pregnant or nursing/breastfeeding.
* Patients with untreated central nervous system metastatic disease.
* Inability to comply with protocol required procedures
* Active, uncontrolled, systemic bacterial, fungal, or viral infections at Screening. NOTE: Oral antibiotics for a controlled infection (e.g., urinary tract infection) are permitted provided that the symptoms are mild and expected to resolve with appropriate treatment at the discretion of the investigator. Subjects on antimicrobial, antifungal, or antiviral prophylaxis are not specifically excluded if all other inclusion/exclusion criteria are met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
To estimate the median progression free survival (mPFS) | From the time of first dose to the occurrence of disease progression (as accessed by mRECIST v1.1) or death due to any cause prior to documented disease progression, up to 2 years..
  mPFS will be summarized with a Kaplan-Meier curve

SECONDARY OUTCOMES:
To determine KIT mutations in tumor tissue and circulating tumor DNA (ctDNA) associated with primary and acquired resistance to combination bezuclastinib and sunitinib. | 1 year
To determine the objective response rate (ORR; complete responses + partial responses) at 16 weeks and total ORR in patients treated with bezuclastinib in combination with sunitinib. | 16 weeks
To determine the clinical benefit rate (complete responses + partial responses + stable disease) at 16 weeks in patients treated with bezuclastinib in combination with sunitinib. | 16 weeks
To estimate the overall survival, including the overall survival rates at year one and year two. | 1 year, 2 year
To describe the adverse event profile of bezuclastinib in combination with sunitinib. | 1 year
To describe patient-reported quality of life outcome measures. | 1 year
  Quality of life will be evaluated using the EORTC-QLQ-C30 with descriptive statistics reported at each timepoint. Changes in quality-of-life measures based on the EORTC-QLQ-C30 will be determined (difference at follow-up and baseline will be summarized). Changes in on-treatment scores compared to baseline will be analyzed to determine patients' perception of their functional status, symptoms, and overall health.

CONTACTS AND LOCATIONS:
Overall Officials: Candace Haddox, MD, Principal Investigator — Dana-Farber Cancer Institute; Andrew Wagner, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Sylvester Comprehensive Cancer Center, University of Miami, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania